CLINICAL TRIAL: NCT06353113
Title: Assessing the Feasibility of a Prenatal Mobile App in Pregnant African American Women: The Mindful Maternity Study
Brief Title: Feasibility of a Prenatal Yoga Mobile App in African American Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jennifer Green, Assistant Professor, San Diego State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS-2023-0254
Record Dates: First submitted 2024-03-04; First posted 2024-04-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Related; Mental Health Issue; Discrimination, Racial; Stress; Depression
Keywords: Feasibility; Yoga; Intervention; Mobile Application; Mindfulness; Physical Activity; Pregnant
MeSH Terms: conditions — Racism; Depression; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Down Dog Prenatal Yoga App (Experimental): Prenatal yoga via Down Dog Prenatal Yoga Mobile App 20 minutes a day, 3 days per week, for 12 weeks.
  Interventions: Behavioral: Down Dog Prenatal Yoga App

INTERVENTIONS:
Behavioral: Down Dog Prenatal Yoga App — The Down Dog prenatal yoga app launched in 2015 and was designed to align with the changes a pregnant body goes through in each trimester. Users can select a practice by trimester, which will offer modification cues to work with a changing body during pregnancy. Users can also customize their experience by boosting things like Heartburn or Pubic Symphysis so they can continue to practice yoga and omit poses that might be uncomfortable. The app also utilizes user feedback, to continuously implement new practices to better their app for user interface.
  All of the prenatal yoga classes were created by a certified and experienced prenatal yoga instructor who has a 200hr yoga certification through Pure Yoga (New York), 80hr prenatal yoga certification through Prenatal Yoga Center (New Yoga), and is Trauma Informed Yoga certified through Exhale to Inhale (New York).

SUMMARY:
The goal of this research is to test if a prenatal yoga app can improve well-being in African American/Black (AA) pregnant women. The main questions it aims to answer are:

1. Is the Down Dog prenatal yoga app feasible for AA pregnant women?
2. How does mental and physical health change after using the Down Dog app for 12-weeks?
3. What cultural adaptations to the Down Dog app are needed?

The study lasts for 12 weeks and participants are asked to:

* do prenatal yoga with the app for at least 20 min/day, three days/week, from home
* wear a Garmin Vivosmart 5 watch daily
* complete four online surveys
* complete an optional virtual interview

This project aims to advance public health by contributing to a broader understanding of how prenatal yoga can support the health and well-being of AA pregnant women and promote optimal maternal and child health outcomes.

DETAILED DESCRIPTION:
Recruitment: The investigators will recruit 50 pregnant African American women from local prenatal clinics, non-profits, and social media.

Eligibility: All interested participants will complete a web-based eligibility screener (~5 minutes). Eligible participants will be asked to schedule a virtual intake appointment to review the consent form with a research team member.

Procedures: Participants must sign an informed consent and complete a Physical Activity Readiness Medical Examination (PARmed-X) for Pregnancy with their healthcare provider before beginning the study. Once participants sign the consent and return a completed PARmed-X form, they will be asked to schedule an in-person enrollment appointment.

During the in-person enrollment appointment, participants will receive a free yoga mat and Garmin Vivosmart 5, and study materials. A research team member will set up the Garmin device for the participant. Participants will be asked to resume normal activities for one week before beginning the intervention and to complete a baseline survey.

After one week of baseline data collection, a research team member will send the participant an email with instructions to download/use the prenatal yoga mobile app and other relevant study materials. Participants will then engage in prenatal yoga using the mobile app for at least 20 min/day, 3 days/week for the next 12 weeks. Participants will receive a mid-intervention survey at 6 weeks, a post-intervention survey at 12 weeks, and will have an opportunity to complete a virtual interview when the study is over. Within 1-2 weeks after the participants' due date, a research team member will send an online birth outcomes survey to collect self-reported birth outcomes.

The baseline, mid-intervention, and post-intervention surveys will ask about mental and physical health and perceptions about using the prenatal mobile app. The optional virtual interview will ask questions related to further understanding the feasibility of the prenatal yoga mobile app and exploring cultural adaptations to improve the app.

ELIGIBILITY:
Inclusion Criteria

Participants will be included in the study if they:

* Are 18-46 years of age (childbearing age)
* Reside in San Diego Metropolitan Area
* Speak English
* Are between 13-28 weeks when intervention starts
* Are primiparous (giving birth for the first time)
* Have a singleton pregnancy (pregnant with only one baby)
* Are yoga naive (<60 min/month for past 6 months)
* Have access to smartphone/mobile device
* Willing to wear a wrist worn fitness tracker for the duration of the study
* Willing to download and use 3 mobile apps for the duration of the study
* Identify as Black or African American
* Return a completed Physical Activity Readiness Medical Examination (PARmed-X) for Pregnancy form (HCP approves participation in prenatal PA program before beginning intervention)

Exclusion Criteria:

* High-risk pregnancy
* Severe psychiatric disorder or substance abuse
* Denial of physical activity participation from physician

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the intervention | Post intervention (12 weeks)
  Assessed using an investigator-developed questionnaire using a 5 point likert scale from strongly agree to strongly disagree. Acceptability benchmark: > 70% of participants report the intervention to be satisfactory, intend to continue using the app, and perceive the app content to be appropriate for pregnancy.
Demand of the intervention | Assessed across 12-week study period
  Assessed by measuring actual use of the mobile app with data analytics provided from Down dog. Demand benchmark: >70% of participants complete at least 75% of their weekly prescribed minutes (i.e., ≥ 45 of 60 minutes per week).
Retention | Assessed across 12-week study period
  Assessed by calculating the proportion of enrolled participants that complete intervention vs withdrawals. Retention benchmark: ≥70% (N=35) complete the intervention.
Ease of recruitment | Assessed at enrollment
  Assessed by evaluating enrollment rate. Recruitment benchmark: >8 participants will be enrolled each month on average.

SECONDARY OUTCOMES:
Discrimination | Baseline, Mid-intervention (6 weeks), and Post-intervention (12 weeks)
  Discrimination will be assessed using the Discrimination in Medical Settings (DMS) Scale. The DMS is a 7-item instrument scored on a 5-point Likert scale (1-never, 2-rarely, 3-sometimes, 4-most of the time, 5-always). Higher scores indicate greater levels of discrimination.
Perceived stress | Baseline, Mid-intervention (6 weeks), and Post-intervention (12 weeks)
  Perceived stress will be measured using the Perceived Stress Scale (PSS-10). The PSS-10 is a 10-item instrument scored on a 5-point Likert scale (0-Never, 1- Almost Never, 2- Sometimes, 3- Fairly Often, 4-Very Often). Higher scores indicate greater levels of perceived stress.
Perinatal Depression | Baseline, Mid-intervention (6 weeks), and Post-intervention (12 weeks)
  Perinatal Depression will be measured using the 10-item Edinburg Postnatal Depression Scale (EPDS). Scores range from 0-30, with "possible depression" defined by a score of 10 or greater.
Self-awareness | Baseline, Mid-intervention (6 weeks), and Post-intervention (12 weeks)
  Self-awareness will be measured using the Self Awareness Outcomes Questionnaire (SAOQ). The SAOQ is a 38-item instrument scored on a 5-point Likert scale (1- Never, 2- Rarely, 3- Occasionally, 4- Frequently, 5- Almost Always). The SAOQ has 4 subscales and the score is determined by calculating the mean of certain items corresponding to each subscale. Higher scores indicate greater frequency of experienced outcomes.
Mindfulness | Baseline, Mid-intervention (6 weeks), and Post-intervention (12 weeks)
  Mindfulness will be measured using the Mindful Attention Awareness Scale (MAAS). The MAAS is a 15-item instrument scored on a 6-point Likert scale (1- Almost Always, 2- Very Frequently, 3- Somewhat Frequently, 4- Somewhat Infrequently, 5- Very Infrequently, 6- Almost Never). Higher scores indicate greater levels of mindfulness.
Subjective physical activity | Baseline, Mid-intervention (6 weeks), and Post-intervention (12 weeks)
  Subjective physical activity will be measured using the Pregnancy Physical Activity Questionnaire (PPAQ). The instrument assesses the approximate amount of time spent in 32 activities including household/caregiving, occupational, sports/exercise, and inactivity during the current trimester. Duration and intensity will be determined using Compendium-based MET values.
Objective physical activity (steps) | Daily for 12 weeks
  The number of steps per day will be measured using the Garmin Vivosmart 5 fitness tracker.
Objective physical activity (intensity) | Daily for 12 weeks
  Intensity of activity will be measured using metabolic equivalents (METs) value via the Garmin Vivosmart 5 fitness tracker.
Cardiac health (heart rate) | Daily for 12 weeks
  Heart rate in beats per minute (BPM) will be measured using the Garmin Vivosmart 5 fitness tracker.
Cardiac health (heart rate variability) | Daily for 12 weeks
  Heart rate variability in milliseconds will be measured using the Garmin Vivosmart 5 fitness tracker.
Cultural adaptations | Post-Intervention (12 weeks)
  Qualitative interviews will be used to explore and identify cultural adaptations relevant for African American pregnant women.
Birth outcomes (gestational age) | Post-delivery (~2 weeks after delivery of baby)
  Self-report survey will be used to assess gestational age (total length of pregnancy in weeks).
Birth outcomes (type of delivery) | Post-delivery (~2 weeks after delivery of baby)
  Self-report survey will be used to assess the type of delivery (e.g., vaginal, planned C-section, unplanned C-section).
Birth outcomes (intervention used for delivery) | Post-delivery (~2 weeks after delivery of baby)
  Self-report survey will be used to assess interventions used for delivery, if applicable, using a list. An intervention can include use of medical treatments or procedures to induce labor or assist with delivery.
Birth outcomes (birth weight) | Post-delivery (~2 weeks after delivery of baby)
  Self-report survey will be used to assess birth weight (weight of baby in pounds + ounces).
Birth outcomes (maternal weight) | Post-delivery (~2 weeks after delivery of baby)
  Self-report survey will be used to assess maternal weight (last known weight before delivery in pounds).
Birth outcomes (pregnancy-related disorders) | Post-delivery (~2 weeks after delivery of baby)
  Self-report survey will be used to assess pregnancy-related disorders, if applicable, using a list. Pregnancy-related disorders could be complications including physical and mental conditions that affect the health of the pregnant or postpartum person, their baby, or both (e.g.,preterm birth, gestational diabetes, preeclampsia, eclampsia, birth injury, postpartum hemorrhage, postpartum hypertension etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Jeni Green, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacDorman MF, Thoma M, Declcerq E, Howell EA. Racial and Ethnic Disparities in Maternal Mortality in the United States Using Enhanced Vital Records, 2016-2017. Am J Public Health. 2021 Sep;111(9):1673-1681. doi: 10.2105/AJPH.2021.306375. Epub 2021 Aug 12. PMID 34383557
- [Background] Ely DM, Driscoll AK. Infant Mortality in the United States, 2020: Data From the Period Linked Birth/Infant Death File. Natl Vital Stat Rep. 2022 Sep;71(5):1-18. PMID 36190428
- [Background] Giurgescu C, Kavanaugh K, Norr KF, Dancy BL, Twigg N, McFarlin BL, Engeland CG, Hennessy MD, White-Traut RC. Stressors, resources, and stress responses in pregnant African American women: a mixed-methods pilot study. J Perinat Neonatal Nurs. 2013 Jan-Mar;27(1):81-96. doi: 10.1097/JPN.0b013e31828363c3. PMID 23360946
- [Background] Knuist M, Bonsel GJ, Zondervan HA, Treffers PE. Risk factors for preeclampsia in nulliparous women in distinct ethnic groups: a prospective cohort study. Obstet Gynecol. 1998 Aug;92(2):174-8. doi: 10.1016/s0029-7844(98)00143-4. PMID 9699746
- [Background] Brown HL, Chireau MV, Jallah Y, Howard D. The "Hispanic paradox": an investigation of racial disparity in pregnancy outcomes at a tertiary care medical center. Am J Obstet Gynecol. 2007 Aug;197(2):197.e1-7; discussion 197.e7-9. doi: 10.1016/j.ajog.2007.04.036. PMID 17689648
- [Background] Dagher RK, Linares DE. A Critical Review on the Complex Interplay between Social Determinants of Health and Maternal and Infant Mortality. Children (Basel). 2022 Mar 10;9(3):394. doi: 10.3390/children9030394. PMID 35327766
- [Background] Larson CP. Poverty during pregnancy: Its effects on child health outcomes. Paediatr Child Health. 2007 Oct;12(8):673-7. doi: 10.1093/pch/12.8.673. PMID 19030445
- [Background] Narendran S, Nagarathna R, Narendran V, Gunasheela S, Nagendra HR. Efficacy of yoga on pregnancy outcome. J Altern Complement Med. 2005 Apr;11(2):237-44. doi: 10.1089/acm.2005.11.237. PMID 15865489
- [Background] Green J, James D, Larkey L, Leiferman J, Buman M, Oh C, Huberty J. A qualitative investigation of a prenatal yoga intervention to prevent excessive gestational weight gain: A thematic analysis of interviews. Complement Ther Clin Pract. 2021 Aug;44:101414. doi: 10.1016/j.ctcp.2021.101414. Epub 2021 May 6. PMID 33989862
- [Background] Battle CL, Uebelacker LA, Magee SR, Sutton KA, Miller IW. Potential for prenatal yoga to serve as an intervention to treat depression during pregnancy. Womens Health Issues. 2015 Mar-Apr;25(2):134-41. doi: 10.1016/j.whi.2014.12.003. PMID 25747520
- [Background] Green J, Neher T, Puzia M, Laird B, Huberty J. Pregnant women's use of a consumer-based meditation mobile app: A descriptive study. Digit Health. 2022 Mar 27;8:20552076221089098. doi: 10.1177/20552076221089098. eCollection 2022 Jan-Dec. PMID 35371532